CLINICAL TRIAL: NCT04873596
Title: Comparison Between Dexmedetomidine and Midazolam Nebulization as Procedural Sedation During Cesarean Delivery Under Spinal Anesthesia in Pre-eclamptic Parturients
Brief Title: Dexmedetomidine and Midazolam Nebulization as Sedation During Cesarean Delivery in Pre-eclampsia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Alshaimaa Abdel Fattah Kamel, principle investigator, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6869
Record Dates: First submitted 2021-04-25; First posted 2021-05-05 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Procedural Sedation
MeSH Terms: interventions — Dexmedetomidine; Midazolam

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nebulized dexmedetomidine (Active Comparator): parturient will receive nebulized 3ug/kg dexmedetomidine diluted in normal saline (0.9%) solution till total volume of nebulized solution will become 5 ml and will be nebulized by a standard hospital jet nebulizer via mouthpiece, with a continuous flow of 100% oxygen at 6 L/min. for 15 minutes, and the treatment will be stopped when the nebulizer will be began to sputter.
  Interventions: Drug: Nebulized dexmedetomidine
- nebulized midazolam (Active Comparator): parturient will receive nebulized 0.2 mg/kg midazolam diluted in normal saline (0.9%) solution till total volume of nebulized solution will become 5 ml and will be nebulized by a standard hospital jet nebulizer via mouthpiece, with a continuous flow of 100% oxygen at 6 L/min. for 15 minutes, and the treatment will be stopped when the nebulizer will be began to sputter.
  Interventions: Drug: Nebulized midazolam

INTERVENTIONS:
Drug: Nebulized dexmedetomidine — parturient will receive nebulized 3ug/kg dexmedetomidine.
  Other Names: precedex
  Arms: nebulized dexmedetomidine
Drug: Nebulized midazolam — parturient will receive nebulized 0.2 mg/kg midazolam.
  Other Names: Dormicum
  Arms: nebulized midazolam

SUMMARY:
Null hypothesis: There is no difference between the effects of nebulization of dexmedetomidine and midazolam as procedural sedation during cesarean delivery under spinal Anesthesia in pre-eclamptic parturients Alternative hypothesis: There is difference between the effects of nebulization of dexmedetomidine and midazolam as procedural sedation during cesarean delivery under spinal anesthesia in pre-eclamptic parturients

DETAILED DESCRIPTION:
Site of study:

This study will be carried out in operating theater of obstetrics at Zagazig University Hospitals.

Withdrawal Criteria: The woman has the right to withdraw from the study at any time without any negative consequence on their medical or surgical treatment plan.

Double -blind randomized clinical trial. All patients will be hospitalized and visited a day before the surgery, full history with physical examination and routine investigation will be done, the nature and complications of the study will be explained in detail to the patient and informed written consent will be obtained from every woman.

ELIGIBILITY:
Inclusion Criteria:

* Age: 21-38 years old.
* Mild and moderate preeclampsia parturient.
* American Society of AnesthesiologistPhysical status II.
* Body Mass Index (BMI) (25-35kg/m²).
* Type of operations: elective cesarean section under spinal anesthesia.
* Written informed consent from the parturient.

Exclusion Criteria:

* Altered mental state.
* Women with known history of allergy to study drugs.
* Women with uncontrolled diabetes mellitus, bleeding, coagulation disorders, advanced hepatic, renal, cardiovascular, respiratory disease and neuropsychiatric disorders.
* Patients receiving anticonvulsants or antidepressants.
* Sever preeclampsia, intrauterine growth restriction or fetal compromise.

Ages: 21 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 94 (Estimated)
Dates: Start 2021-05-15 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Chane in the level of sedation | at 0 minute (immediately after nebulization) , 5 minutes then every 15 minutes intraoperative
  Change in the level of sedation will be assessed using Ramasy Sedation Assessment Scale
  Ramsay Sedation Scale
  1= Patient is anxious and agitated or restless, or both 3= Patient responds to commands only 4= Patient exhibits brisk response to light glabellar tap or loud auditory stimulus 5= Patient exhibits a sluggish response to light glabellar tap or loud auditory stimulus 6= Patient exhibits no response

SECONDARY OUTCOMES:
The discharge time from Post Anesthesia Care Unite (PACU) . | up to 30 minutes postoperative
  The discharge time from Post Anesthesia Care Unite (PACU) in minutes when achieving modified Aldrete Score 9.
  Modified Aldert Score.
  Activity, able to move, voluntarily or on command 4 extremities = 2 2 extremities = 1 No = 0
  Breathing Able to breathe deeply & cough freely= 2 Dyspnea, shallow or limited breathing =1 Apnea= 0
  Consciousness Fully awake = 2 Arousable on calling = 1 Unresponsive = 0 Circulation (BP) ±20% of pre-anesthesia level= 2
  * 20% to 49% of pre-anesthesia level= 1
  * 50% of pre-anesthesia level= 0
  SPO2 Maintains SpO2 >92% in ambient air= 2 Maintain SpO2 >90% with O2 = 1 Maintain SpO2 <90% with O2 = 0
Maternal satisfaction with procedure | up to 24hour postoperative
  Maternal satisfaction with procedure using a 5-point numerical rating scale. 0= Extremely dissatisfied
  1. Dissatisfied
  2. Neutral
  3. Satisfied
  4. Extremely satisfied
APGAR score | at 1 and 5 min after delivery
  APGAR score at 1 and 5 min after delivery APGAR score (13). Indicator Score 0 Score 1 Score 2 Activity (muscle tone) Limp; no movement Some flexion of arms and legs Active motion Pulse (heart rate) No heart rate Fewer than 100 beats per minute At least 100 beats per minute Grimace (reflex response) No response to airways being suctioned Grimace during suctioning Grimace and pull away, cough, or sneeze during suctioning Appearance (color) The baby's whole body is completely bluish-gray or pale Good color in body with bluish hands or feet Good color all over Respiration (breathing) Not breathing Weak cry; may sound like whimpering, slow or irregular breathing Good, strong cry; normal rate and effort of breathing
  Total Score: 3 and below require immediate resuscitation 4 to 7 may require resuscitative measures 7 to 10 is considered normal
Heart rate | Baseline, at 0 minute (after nebulization), 5 minutes then every 10 minutes intraoperative.
  heart rate in beat/ minute
Mean arterial blood pressure | Baseline, at 0 minute (after nebulization), 5 minutes then every 10 minutes intraoperative.
  Mean arterial blood pressure in mmHg
Oxygen saturation | Baseline, at 0 minute (after nebulization), 5 minutes then every 10 minutes intraoperative.
  Oxygen saturation by pulse oximetry.

CONTACTS AND LOCATIONS:
Overall Officials: Alshaimaa Kamel, M.D, Principal Investigator — Zagazig University, Faculty of human medicine
Locations (1):
- Zagazig University, Faculty of medicine, Zagazig, Egypt